CLINICAL TRIAL: NCT01974596
Title: THE EFFECT OF ORALLY ADMINISTERED PROBIOTIC LACTOBACILLUS REUTERI-CONTAINING TABLETS IN PERI-IMPLANT MUCOSITIS: A RANDOMIZED CLINICAL TRIAL
Brief Title: Use of Probiotics in Oral Health of Patients With Dental Implants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Antonio Juan Flichy Fernández, DDS, Colaborator University of Valencia, University of Valencia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Probiotics
Record Dates: First submitted 2013-10-15; First posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Mucositis
Keywords: Dental implants; Probiotics; Lactobacillus reuteri; Periimplant mucositis; Cytokines; Bacterial load
MeSH Terms: conditions — Mucositis | interventions — Probiotics; Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Probiotic Lactobacillus reuteri Vs Placebo (Experimental): patients with full arch with dental implant received a tablet of Lactobacillus reuteri every day during 28 days, and after a wash-up, the same patients receive a tablet of placebo every day during 28 days
  Interventions: Dietary Supplement: Probiotic tablets of Lactobacillus reuteri; Dietary Supplement: Placebo tablets

INTERVENTIONS:
Dietary Supplement: Probiotic tablets of Lactobacillus reuteri
  Other Names: strains of Lactobacillus reuteri ATCC PTA 5289 - 100 million; Strains of Lactobacillus reuteri DSM 17938 - 100 million
Dietary Supplement: Placebo tablets
  Other Names: Placebo tablets with same visually aspect, flavour and texture than the probiotic but without probiotic strains

SUMMARY:
The aim of this study was evaluate the effects of the oral probiotic Lactobacillus reuteri Prodentis upon the peri-implant health of edentulous patients with dental implants and peri-implant mucositis, establishing comparisons versus implants without peri-implant disease. The hypothesis of the study is that using these probiotics are going to improve the periimplant health.

DETAILED DESCRIPTION:
A double-blind, placebo-controlled, prospective cross-over study was made. All the patients were edentulous and were divided into two groups: A) with no peri-implant disease; B) with peri-implant mucositis affecting one or more implants. Patients with peri-implantitis were excluded. All patients in both groups initially received the oral probiotic Lactobacillus reuteri Prodentis, followed by placebo. Only the supervisor of the study knew this information; clinical examiner and patients were blind. Were studied: crevicular fluid volume, modified plaque index, probing depth, modified gingival index, and concentrations of interleukin 1β, interleukin 6 and interleukin 8, and Bacterial load.

ELIGIBILITY:
Inclusion Criteria:

* Totally edentulous patients subjected to dental implant rehabilitation in one or both arches
* Prosthetic restoration in function for at least 24 months
* Healthy individuals without known disease

Exclusion Criteria:

* Patients receiving any kind of local or systemic decontamination treatment of the oral cavity (e.g., antibiotics or rinses) in the last 3 months, or periodontal treatment in the last 6 months
* Uncontrolled periodontal disease
* Patients with immune deficiencies, diabetes, rheumatoid disease, head and neck radiotherapy, bisphosphonate treatment, chemotherapy or anticoagulation
* Patients with dental implants presenting intraoral exposure of the rough portion of any implant
* Smokers
* Incomplete protocols due to a lack of patient cooperation: a) failure to follow the treatment instructions; b) failure to report to the visit after one month of follow-up
* Failure to provide informed consent to participation the study
* Patients presenting at least one implant with peri-implantitis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Evidence in reduction of plaque index | 28 days using one probiotic tablet/day
  The Mombelli clasification was used to evaluate the reduction of bacterial plaque. 0: No bacterial plaque; 1: presence of bacterial plaque but not visually; 2: 1/3 part of the implant with bacterial plaque; 3: 2/3 parts or more of the implant with bacterial plaque

SECONDARY OUTCOMES:
Evidence in reduction of bleeding around implants | 28 days using probiotic tablet/day
  The Mombelli classification was used to evaluate the reduction of bleeding around implants: 0: no bleeding; 1: a point of bleeding; 2)a line of bleeding; 3: much bleeding
Evidence in reduction of probing depth | 28 days using one probiotic tablet/day
  Was measured in reduction of millimeters of the depth of the implant with a millimeter probe.
Evidence in reduction Interleukin 1β concentration | 28 days using one probiotic tablet/day
  concentration measured in picograms/milliliter (pg/ml)
Evidence in reduction Interleukin 6 concentration | 28 days using one probiotic tablet/day
  concentration measured in picograms/milliliter (pg/ml)
Evidence in reduction Interleukin 8 concentration | 28 days using one probiotic tablet/day
  concentration measured in picograms/milliliter (pg/ml)

OTHER OUTCOMES:
Evidence of reduction of Total Bacterial Load studied | 28 days using probiotic tablets/day
  Where evaluate Aggregatibacter and red complex of socransky

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral Surgery, University of Valencia, Valencia, Valencia, Spain